CLINICAL TRIAL: NCT05002231
Title: A Phase 1, Open-Label, 3-Period, Randomized, Single-Dose, Crossover Study to Assess the Relative Bioavailability and the Effect of Food on the Pharmacokinetics of a New 15 mg Tablet of Losmapimod Versus the Current 7.5 mg Tablet
Brief Title: Relative Bioavailability and Food Effect Study of Losmapimod 15 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1821-CLP-101
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Healthy Adult Subjects
Keywords: Healthy Adult Subjects
MeSH Terms: interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide; Tablets

STUDY DESIGN:
Intervention Model Description: Open-label, 3-period, 6-sequence, randomized, single-dose, crossover study designed to assess the relative bioavailability of a 15 mg tablet of losmapimod versus two 7.5 mg tablets of losmapimod under fasted conditions and to assess the effect of food on the pharmacokinetics of a 15 mg tablet of losmapimod under fasted and fed conditions
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, single-dose, cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Losmapimod 15 mg oral tablet in healthy subjects (Treatment Regimen A) (Experimental): Subjects will be randomized to 1 of 6 treatment sequences to receive one 15 mg tablet of losmapimod administered orally under fasted conditions. Subjects will fast overnight (nothing to eat or drink except water) for at least 10 hours before each study drug administration. Subjects will remain fasted for 4 hours after dosing with study drug. Washout period of 48 hours between dosing.
  Interventions: Drug: Losmapimod 15 mg oral tablet
- Losmapimod two 7.5 mg oral tablets in healthy subjects (Treatment Regimen B) (Experimental): Subjects will be randomized to 1 of 6 treatment sequences to receive two 7.5 mg tablets of losmapimod administered orally under fasted conditions. Subjects will fast overnight (nothing to eat or drink except water) for at least 10 hours before each study drug administration. Subjects will remain fasted for 4 hours after dosing with study drug. Washout period of 48 hours between dosing.
  Interventions: Drug: Losmapimod two 7.5 mg oral tablets
- Losmapimod one 15 mg oral tablet in healthy subjects (Treatment Regimen C) (Experimental): Subjects will be randomized to 1 of 6 treatment sequences to receive one 15 mg tablet of losmapimod administered orally under fed conditions. Subjects will fast overnight (nothing to eat or drink except water) for at least 10 hours before breakfast and will receive a high-fat breakfast approximately 30 minutes before dose administration. Subjects must consume the meal within 25 minutes or less. Washout period of 48 hours between dosing.
  Interventions: Drug: Losmapimod one 15 mg oral tablet

INTERVENTIONS:
Drug: Losmapimod 15 mg oral tablet — Subjects will receive one losmapimod 15 mg tablet by mouth under fasted conditions.
  Arms: Losmapimod 15 mg oral tablet in healthy subjects (Treatment Regimen A)
Drug: Losmapimod two 7.5 mg oral tablets — Subjects will receive two losmapimod 7.5 mg tablets by mouth under fasted conditions.
  Arms: Losmapimod two 7.5 mg oral tablets in healthy subjects (Treatment Regimen B)
Drug: Losmapimod one 15 mg oral tablet — Subjects will receive one losmapimod 15 mg tablet by mouth under fed conditions.
  Arms: Losmapimod one 15 mg oral tablet in healthy subjects (Treatment Regimen C)

SUMMARY:
This is a study to assess the relative bioavailability and the effect of food on the pharmacokinetics of a new 15 mg tablet formulation of losmapimod

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, 3-period, 6-sequence, randomized, single-dose, crossover study designed to assess the relative bioavailability of a 15 mg tablet of losmapimod versus two 7.5 mg tablets of losmapimod under fasted conditions and to assess the effect of food on the pharmacokinetics of a 15 mg tablet of losmapimod under fasted and fed conditions in 18 healthy subjects.

The study will consist of a screening period, 3 treatment periods with a single dose of study drug per treatment period, a 48-hour washout period between dosing, and an end of study visit. Subjects will be randomly assigned to receive 1 of 6 treatment sequences (3 subjects per treatment sequence) prior to dosing on Day 1 of Period 1.

The primary endpoint of the study is to assess the relative bioavailability and the effect of food on the pharmacokinetics of a new 15 mg tablet formulation of losmapimod. Secondary endpoints include assessing the safety and tolerability and evaluating target engagement in the blood of a new 15 mg tablet formulation of losmapimod in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, 18 to 65 years of age, inclusive, at screening.
2. Body mass index 18 to 30 kg/m2, inclusive, at screening with a minimum weight of 50 kg.
3. Good general health, based upon the opinion of the investigator as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at screening.
4. Willingness of men and women of reproductive potential must agree to use 2 effective and acceptable methods of contraception throughout study participation until 90 days after last dose of study drug. Female subjects must have a negative pregnancy test at screening and before the first dose of study drug.
5. Willing and able to comply with all protocol requirements.
6. The subject is able to provide written informed consent.

Exclusion Criteria:

1. History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include, but is not limited to, history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; history or presence of clinically significant pathology; clinically significant history of mental disease; and history of cancer, except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ (all 3 with no recurrence for the last 5 years).
2. History of febrile illness within 5 days before the first dose of study drug.
3. Current clinically significant liver or kidney dysfunction.
4. Acute or chronic history of liver disease or current alanine aminotransferase elevation >1.5 × upper limit of normal (ULN) and/or total bilirubin >1.5 × ULN at screening.
5. Positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
6. Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy, or other gastrointestinal tract surgery, except appendectomy).
7. Standard 12 lead ECG demonstrating QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 msec for male subjects and QTcF >470 msec for female subjects at screening. If QTcF exceeds 450 msec for males or 470 msec for females, the ECG will be repeated 2 more times, and the average of the 3 QTcF values will be used to determine the subject's eligibility.
8. History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s) or history or evidence of abnormal ECGs that, in the opinion of the investigator or medical monitor, would preclude the subject's participation in the study.
9. Blood or blood product (e.g., plasma/serum) donation (of approximately 1 pint [500 mL] or more) or has any significant loss of blood within 3 months (males) or 4 months (females) prior to screening or intention to donate blood or blood products during the study as determined by the investigator.
10. History of abuse of addictive substances such as drug abuse, or regular user of sedatives, hypnotics, tranquilizers, or any other addictive agent within 6 months prior to screening.
11. History of regular alcohol consumption within 6 months prior to screening defined as an average weekly intake of greater than 21 units. One unit is equivalent to approximately half pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits.
12. History of demonstrating an excess in xanthine consumption (more than 8 cups of coffee or equivalent per day).
13. Received study drug in another investigational study within 30 days of dosing.
14. Received the coronavirus disease 2019 (COVID-19) vaccine within 14 days before Day 1, or subjects who plan to receive a COVID-19 vaccine at any time during the study, including during the follow up period or has tested positive for COVID 19 within 3 months prior to screening.
15. Use of any medication (prescription or over-the-counter) within 14 days of study drug administration, or use of herbal supplements, dietary supplements, or multivitamins within 7 days of study drug administration or less than five half-lives (whichever is longer), with the exception of contraceptives, hormonal replacement therapies, and acetaminophen (up to 3 grams per day). Other exceptions will only be made if the rationale is clearly documented by the investigator.
16. History of sensitivity to the study drug, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicated their participation.
17. Female subjects who are lactating or pregnant as determined by positive serum human chorionic gonadotropin test at screening or on Day -1.
18. Subject is mentally or legally incapacitated.
19. Abnormal laboratory results indicative of any significant medical disease that, in the opinion of the investigator, would preclude the subject's participation in the study at screening or prior to first dose of study drug.
20. Subject, or close relative of the subject, is the investigator or a sub-investigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study at that study site.
21. Subject smokes cigarettes (or equivalent including vaping) and/or has used nicotine based products within 14 days prior to screening.
22. Positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or on Day -1.
23. Consumption of grapefruit or grapefruit juice, Seville orange or Seville orange containing products (e.g., marmalade), or alcohol-, caffeine-, or xanthine containing products within 48 hours before the first dose of study drug.
24. Plans for hospitalization, surgery, or other major procedures during the study duration between the screening visit and Day -1.
25. In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of Losmapimod | Treatment Regimen A: Days 1 and 2
  To assess the bioavailability of losmapimod (1 x 15 mg tablet) (test) versus losmapimod tablets (2 x 7.5 mg tablets) (reference), blood samples will be collected under fasted conditions to measure the plasma concentration of losmapimod at specified timepoints by liquid chromatography with tandem mass spectrometry.
Plasma Concentrations of Losmapimod | Treatment Regimen B: Days 1 and 2
  To assess the bioavailability of losmapimod (1 x 15 mg tablet) (test) versus losmapimod tablets (2 x 7.5 mg tablets) (reference), blood samples will be collected under fasted conditions to measure the plasma concentration of losmapimod at specified timepoints by liquid chromatography with tandem mass spectrometry.
Food Effect of Losmapimod | Treatment Regimen A: Days 1 and 2
  To assess the effect of food on the pharmacokinetics of losmapimod test versus reference, blood samples will be collected under fasted conditions to measure the plasma concentration of losmapimod at specified timepoints by liquid chromatography with tandem mass spectrometry.
Food Effect of Losmapimod | Treatment Regimen Part C: Days 1 and 2
  To assess the effect of food on the pharmacokinetics of losmapimod, blood samples will be collected after a high fat meal to measure the plasma concentration of losmapimod at specified timepoints by liquid chromatography with tandem mass spectrometry.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events | Up to approximately 4 weeks of monitoring
  To evaluate the safety and tolerability of losmapimod 15 mg in healthy adult subjects based on the frequency of adverse events (AEs), frequency of serious adverse events (SAEs), and clinically significant laboratory test results, electrocardiograms (ECGs), vital signs and physical examination findings.
Target Engagement in Blood | Treatment Regimen A: Day 1
  Change from baseline in the ratio of phosphor-HSP27/total-HSP27 in sorbitol-stimulated whole blood lysate will be evaluated by enzyme linked immunosorbent assay (ELISA).
Target Engagement in Blood | Treatment Regimen B: Day 1
  Change from baseline in the ratio of phosphor-HSP27/total-HSP27 in sorbitol-stimulated whole blood lysate will be evaluated by enzyme linked immunosorbent assay (ELISA).
Target Engagement in Blood | Treatment Regimen C: Day 1
  Change from baseline in the ratio of phosphor-HSP27/total-HSP27 in sorbitol-stimulated whole blood lysate will be evaluated by enzyme linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mellion, MD, Study Director — Fulcrum Therapeutics
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour AM, Sarov-Blat L, Cai G, Fossler MJ, Sprecher DL, Graggaber J, McGeoch AT, Maison J, Cheriyan J. Safety, tolerability, pharmacokinetics and pharmacodynamics of losmapimod following a single intravenous or oral dose in healthy volunteers. Br J Clin Pharmacol. 2013 Jul;76(1):99-106. doi: 10.1111/bcp.12063. PMID 23215699
- [Background] Mellion ML, Ronco L, Berends CL, Pagan L, Brooks S, van Esdonk MJ, van Brummelen EMJ, Odueyungbo A, Thompson LA, Hage M, Badrising UA, Raines S, Tracewell WG, van Engelen B, Cadavid D, Groeneveld GJ. Phase 1 clinical trial of losmapimod in facioscapulohumeral dystrophy: Safety, tolerability, pharmacokinetics, and target engagement. Br J Clin Pharmacol. 2021 Dec;87(12):4658-4669. doi: 10.1111/bcp.14884. Epub 2021 May 14. PMID 33931884